CLINICAL TRIAL: NCT04352335
Title: Change in Neutrophil to Lymphocyte Ratio (NLR) and Survival Among Advanced Lung Cancer Patients Receiving Immune Checkpoint Inhibitors With Immunomodulator: a Retrospective Study
Brief Title: Change in NLR and Survival Among Advanced Lung Cancer Patients Receiving ICIs With Immunomodulator
Status: Completed | Type: Observational
Sponsor: Chung Shan Medical University (Other)
Responsible Party: Principal Investigator, LJ Hwu, Attending physician, Chung Shan Medical University
Other Study IDs: CSMUH02-NLR
Record Dates: First submitted 2020-04-16; First posted 2020-04-20 (Actual); Last update posted 2020-07-02 (Actual); Status verified 2020-06

CONDITIONS: Advanced Lung Cancer
Keywords: neutrophil to lymphocyte ratio (NLR); immunomodulator

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cohort 1：ICI treatment with immunomodulator: Lung cancer patients received immunological checkpoint inhibitors (ICIs) and any immunomodulatory drugs.
- Cohort 2：ICI treatment without immunomodulator: Lung cancer patients received immunological checkpoint inhibitors (ICIs).

SUMMARY:
The main objective of this study is to evaluate the change of neutrophil to lymphocyte ratio (NLR) after 6-week treatment of immune checkpoint inhibitors (ICIs) with or without immunomodulatory drugs and recognize the effect of post-treatment NLR and overall survival in advanced lung cancer patients by retrospective review.

DETAILED DESCRIPTION:
In recent years, the therapeutic strategies for lung cancer have been enriched with small molecular targeted therapy and immunotherapy. In this retrospective study, we will observe the change in NLR and explore its possible association with survival among advanced lung cancer patients receiving Immune checkpoint inhibitors (ICIs) with and without such immuno-modulator, Astragalus Polysaccharide Injection. It can be used to understand the relationship between NLR values and the survival rate of lung cancer patients after ICIs treatment. Physicians can refer to this result to give patients the suitable treatment recommendations.

ELIGIBILITY:
Inclusion Criteria

* Aged 20 years and older.
* Patients who have been given a diagnosis of lung cancer.
* Previously advanced lung cancer patients first treated with ICIs from Oct 1, 2015 to Oct 31, 2019.

Exclusion Criteria

* Patients who have no hematological laboratory data available at baseline (within 3 days prior to ICI treatment) and the 6th week (± 2 weeks) after ICI treatment initiation.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with lung cancer undergoing ICIs with or without immunomodulatory drug
Sampling Method: Non-Probability Sample
Enrollment: 53 (Actual)
Dates: Start 2020-04-14 (Actual); Primary Completion 2020-07-01 (Actual); Study Completion 2020-07-01 (Actual)

PRIMARY OUTCOMES:
Neutrophil to lymphocyte ratio (NLR) | Baseline, 4~8 week

SECONDARY OUTCOMES:
Overall Survival (OS) | 4 years

CONTACTS AND LOCATIONS:
Overall Officials: Shih-Ming TSAI, M.D., Ph.D., Principal Investigator — Chung Shan Medical University
Locations (1):
- Chung Shan Medical University Hospital, Taichung, Taiwan

IPD SHARING:
Plan to Share IPD: No